CLINICAL TRIAL: NCT00327678
Title: Young Adult With Acute Lymphoblastic Leukemia (ALL) : a Multicentric Protocol. GRAALL 2005 : T ALL or B ALL Non Ph GRAALL 2005 R : B ALL Non Ph CD20+ GRAAPH 2005 : ALL Ph
Brief Title: Treatment of Acute Lymphoblastic Leukemia (ALL) in Younger Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Group for Research in Adult Acute Lymphoblastic Leukemia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRAALL 2005
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-03

CONDITIONS: Leukemia, Lymphocytic
Keywords: ALL,; young patients,; chemotherapy,; Mabtera,; Imatinib,; allogeneic transplant
MeSH Terms: conditions — Leukemia, Lymphoid | interventions — Rituximab; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rituximab
Drug: Imatinib Mesylate

SUMMARY:
This study is a multicenter trial of treatment for young ALL patients. All ALL patients will receive the same steroid pre-phase in order to evaluate sensitivity or resistance. Then, patients will be included into 3 specific trials according to biological features (immunophenotype, cytogenetics, and molecular biology).

Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL) 2005:

* T ALL or B ALL non Ph (N=810 patients planned).
* GRAALL 2005 R: B ALL non Ph CD20+ (N=220 patients planned).
* GRAAPH 2005: ALL Ph+ (N=270 patients planned)

DETAILED DESCRIPTION:
GRAALL 2005: T ALL or B ALL non Ph

Randomization between standard versus intensified cyclophosphamide administration during a 4-drug, 4 week chemotherapy and late intensification.

(N=810 patients planned)

GRAALL 2005 R: B ALL non Ph CD20+

Randomization between standard versus intensified cyclophosphamide administration during a 4-drug, 4 week chemotherapy and late intensification.

Randomization between Mabthera (rituximab) or no Mabthera during all induction and consolidation courses.(N=220 patients planned)

Allogenic transplantation will be performed depending on unfavourable risk factors.

GRAAPH 2005: ALL Ph

Randomization between an imatinib-based induction and a chemotherapy + imatinib induction. (N=270 patients planned)

Allogenic transplantation will be systematically performed in the presence of related or unrelated donors.

Autologous transplantation could be performed in the absence of a donor in case of Molecular Residual Disease (MRD) ≤ 10-4.

Consolidation therapy will be performed in the absence of a donor in case of MRD > 10-4.

ELIGIBILITY:
Inclusion Criteria:

* 18-59 years
* ALL newly diagnosed (blast < 20%)
* Central Nervous System (CNS) positive or negative
* Signed written informed consent
* For GRAAPH trial only: t(9;22) or BCR- ABL positive

Exclusion Criteria:

* Lymphoblastic lymphoma
* ALL 3
* Chronic myeloid leukemia
* Severe organ condition

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1080 (Actual)
Dates: Start 2006-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Event free survival for all patients | January 2014
GRAAPH: Percentage of patients with minimum residual disease (MRD) < 10-4 after induction and/or consolidation (= salvage) | January 2014

SECONDARY OUTCOMES:
CR in 1 or 2 courses | January 2014
Death in induction | January 2014
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | January 2014
Death in first CR | January 2014
Relapse | January 2014
Relapse free survival | January 2014
Overall Survival | January 2014

CONTACTS AND LOCATIONS:
Overall Officials: HERVE DOMBRET, MD, PHD, Study Chair — GRAALL Group
Locations (1):
- Group for Research in Adult Acute Lymphoblastic Leukemia - GRAALL -, Lyon, France

REFERENCES:
- [Derived] Delafoy M, Bonnet MF, Lengline E, Cieslak A, Touzart A, Balducci E, Simonin M, Lheritier V, Dourthe ME, Heid-Picard B, Latour S, Dombret H, Rousselot P, Baruchel A, Boissel N, Andrieu GP, Asnafi V. LEF1 intragenic deletion induces a dominant-negative isoform and unveils a Wnt/beta-catenin vulnerability in T-ALL. Blood. 2025 Dec 18;146(25):3036-3049. doi: 10.1182/blood.2025030161. PMID 40857670
- [Derived] Simonin M, Vasseur L, Lengline E, Lhermitte L, Cabannes-Hamy A, Balsat M, Schmidt A, Dourthe ME, Touzart A, Graux C, Grardel N, Cayuela JM, Arnoux I, Gandemer V, Huguet F, Ducassou S, Lheritier V, Chalandon Y, Ifrah N, Dombret H, Macintyre E, Petit A, Rousselot P, Lambert J, Baruchel A, Boissel N, Asnafi V. NGS-based stratification refines the risk stratification in T-ALL and identifies a very-high-risk subgroup of patients. Blood. 2024 Oct 10;144(15):1570-1580. doi: 10.1182/blood.2023023754. PMID 38848537
- [Derived] Balducci E, Simonin M, Duployez N, Steimle T, Dourthe ME, Villarese P, Ducassou S, Arnoux I, Cayuela JM, Balsat M, Courtois L, Andrieu G, Touzart A, Huguet F, Petit A, Ifrah N, Dombret H, Baruchel A, Macintyre E, Preudhomme C, Boissel N, Asnafi V. Genomic imbalance analysis provides new insight into prognostic factors in adult and pediatric T-ALL. Blood. 2024 Aug 29;144(9):988-1000. doi: 10.1182/blood.2023022154. PMID 38518104
- [Derived] Orvain C, Balsat M, Tavernier E, Marolleau JP, Pabst T, Chevallier P, de Gunzburg N, Cacheux V, Huguet F, Chantepie S, Caillot D, Chalandon Y, Frayfer J, Bonmati C, Lheritier V, Ifrah N, Dombret H, Boissel N, Hunault-Berger M. Thromboembolism prophylaxis in adult patients with acute lymphoblastic leukemia treated in the GRAALL-2005 study. Blood. 2020 Jul 16;136(3):328-338. doi: 10.1182/blood.2020004919. PMID 32321172
- [Derived] Touzart A, Boissel N, Belhocine M, Smith C, Graux C, Latiri M, Lhermitte L, Mathieu EL, Huguet F, Lamant L, Ferrier P, Ifrah N, Macintyre E, Dombret H, Asnafi V, Spicuglia S. Low level CpG island promoter methylation predicts a poor outcome in adult T-cell acute lymphoblastic leukemia. Haematologica. 2020 Jun;105(6):1575-1581. doi: 10.3324/haematol.2019.223677. Epub 2019 Sep 19. PMID 31537687
- [Derived] Bond J, Touzart A, Lepretre S, Graux C, Bargetzi M, Lhermitte L, Hypolite G, Leguay T, Hicheri Y, Guillerm G, Bilger K, Lheritier V, Hunault M, Huguet F, Chalandon Y, Ifrah N, Macintyre E, Dombret H, Asnafi V, Boissel N. DNMT3A mutation is associated with increased age and adverse outcome in adult T-cell acute lymphoblastic leukemia. Haematologica. 2019 Aug;104(8):1617-1625. doi: 10.3324/haematol.2018.197848. Epub 2019 Jan 17. PMID 30655366
- [Derived] Huguet F, Chevret S, Leguay T, Thomas X, Boissel N, Escoffre-Barbe M, Chevallier P, Hunault M, Vey N, Bonmati C, Lepretre S, Marolleau JP, Pabst T, Rousselot P, Buzyn A, Cahn JY, Lheritier V, Bene MC, Asnafi V, Delabesse E, Macintyre E, Chalandon Y, Ifrah N, Dombret H; Group of Research on Adult ALL (GRAALL). Intensified Therapy of Acute Lymphoblastic Leukemia in Adults: Report of the Randomized GRAALL-2005 Clinical Trial. J Clin Oncol. 2018 Aug 20;36(24):2514-2523. doi: 10.1200/JCO.2017.76.8192. Epub 2018 Jun 4. PMID 29863974
- [Derived] Maury S, Chevret S, Thomas X, Heim D, Leguay T, Huguet F, Chevallier P, Hunault M, Boissel N, Escoffre-Barbe M, Hess U, Vey N, Pignon JM, Braun T, Marolleau JP, Cahn JY, Chalandon Y, Lheritier V, Beldjord K, Bene MC, Ifrah N, Dombret H; for GRAALL. Rituximab in B-Lineage Adult Acute Lymphoblastic Leukemia. N Engl J Med. 2016 Sep 15;375(11):1044-53. doi: 10.1056/NEJMoa1605085. PMID 27626518
- [Derived] Bond J, Marchand T, Touzart A, Cieslak A, Trinquand A, Sutton L, Radford-Weiss I, Lhermitte L, Spicuglia S, Dombret H, Macintyre E, Ifrah N, Hamel JF, Asnafi V. An early thymic precursor phenotype predicts outcome exclusively in HOXA-overexpressing adult T-cell acute lymphoblastic leukemia: a Group for Research in Adult Acute Lymphoblastic Leukemia study. Haematologica. 2016 Jun;101(6):732-40. doi: 10.3324/haematol.2015.141218. Epub 2016 Mar 4. PMID 26944475
- [Derived] Chalandon Y, Thomas X, Hayette S, Cayuela JM, Abbal C, Huguet F, Raffoux E, Leguay T, Rousselot P, Lepretre S, Escoffre-Barbe M, Maury S, Berthon C, Tavernier E, Lambert JF, Lafage-Pochitaloff M, Lheritier V, Chevret S, Ifrah N, Dombret H; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL). Randomized study of reduced-intensity chemotherapy combined with imatinib in adults with Ph-positive acute lymphoblastic leukemia. Blood. 2015 Jun 11;125(24):3711-9. doi: 10.1182/blood-2015-02-627935. Epub 2015 Apr 15. PMID 25878120
- [Derived] Chien WW, Catallo R, Chebel A, Baranger L, Thomas X, Bene MC, Gerland LM, Schmidt A, Beldjord K, Klein N, Escoffre-Barbe M, Leguay T, Huguet F, Larosa F, Hayette S, Plesa A, Ifrah N, Dombret H, Salles G, Chassevent A, Ffrench M. The p16(INK4A)/pRb pathway and telomerase activity define a subgroup of Ph+ adult Acute Lymphoblastic Leukemia associated with inferior outcome. Leuk Res. 2015 Apr;39(4):453-61. doi: 10.1016/j.leukres.2015.01.008. Epub 2015 Jan 25. PMID 25675863
- [Derived] Dhedin N, Huynh A, Maury S, Tabrizi R, Beldjord K, Asnafi V, Thomas X, Chevallier P, Nguyen S, Coiteux V, Bourhis JH, Hichri Y, Escoffre-Barbe M, Reman O, Graux C, Chalandon Y, Blaise D, Schanz U, Lheritier V, Cahn JY, Dombret H, Ifrah N; GRAALL group. Role of allogeneic stem cell transplantation in adult patients with Ph-negative acute lymphoblastic leukemia. Blood. 2015 Apr 16;125(16):2486-96; quiz 2586. doi: 10.1182/blood-2014-09-599894. Epub 2015 Jan 13. PMID 25587040
- [Derived] Beldjord K, Chevret S, Asnafi V, Huguet F, Boulland ML, Leguay T, Thomas X, Cayuela JM, Grardel N, Chalandon Y, Boissel N, Schaefer B, Delabesse E, Cave H, Chevallier P, Buzyn A, Fest T, Reman O, Vernant JP, Lheritier V, Bene MC, Lafage M, Macintyre E, Ifrah N, Dombret H; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL). Oncogenetics and minimal residual disease are independent outcome predictors in adult patients with acute lymphoblastic leukemia. Blood. 2014 Jun 12;123(24):3739-49. doi: 10.1182/blood-2014-01-547695. Epub 2014 Apr 16. PMID 24740809
- [Derived] Trinquand A, Tanguy-Schmidt A, Ben Abdelali R, Lambert J, Beldjord K, Lengline E, De Gunzburg N, Payet-Bornet D, Lhermitte L, Mossafa H, Lheritier V, Bond J, Huguet F, Buzyn A, Leguay T, Cahn JY, Thomas X, Chalandon Y, Delannoy A, Bonmati C, Maury S, Nadel B, Macintyre E, Ifrah N, Dombret H, Asnafi V. Toward a NOTCH1/FBXW7/RAS/PTEN-based oncogenetic risk classification of adult T-cell acute lymphoblastic leukemia: a Group for Research in Adult Acute Lymphoblastic Leukemia study. J Clin Oncol. 2013 Dec 1;31(34):4333-42. doi: 10.1200/JCO.2012.48.5292. Epub 2013 Oct 28. PMID 24166518
- [Derived] Ben Abdelali R, Asnafi V, Petit A, Micol JB, Callens C, Villarese P, Delabesse E, Reman O, Lepretre S, Cahn JY, Guillerm G, Berthon C, Gardin C, Corront B, Leguay T, Bene MC, Ifrah N, Leverger G, Dombret H, Macintyre E. The prognosis of CALM-AF10-positive adult T-cell acute lymphoblastic leukemias depends on the stage of maturation arrest. Haematologica. 2013 Nov;98(11):1711-7. doi: 10.3324/haematol.2013.086082. Epub 2013 Jul 5. PMID 23831922